CLINICAL TRIAL: NCT04457284
Title: A Phase II Study of Temozolomide, Cisplatin and Nivolumab in MMR-Proficient Colorectal Cancer
Brief Title: Temozolomide, Cisplatin, and Nivolumab in People With Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-202
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Adenocarcinoma
Keywords: Temozolomide; Cisplatin,; Nivolumab; 20-202
MeSH Terms: interventions — Temozolomide; Cisplatin; Nivolumab

STUDY DESIGN:
Intervention Model Description: This will be a two-stage design, single arm, phase II study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- temozolomide, cisplatin and nivolumab (Experimental): Subjects will receive oral TMZ at 150-200 mg/m2 day 1 to 5 every 4 weeks, cisplatin via IV infusion at 40 mg/m2 every two weeks (Q2W), and nivolumab via IV infusion at 480 mg every four weeks (Q4W).
  Interventions: Drug: Temozolomide (TMZ); Drug: Cisplatin; Drug: Nivolumab

INTERVENTIONS:
Drug: Temozolomide (TMZ) — TMZ 150 mg/m2 Day 1 - 5 Q4W PO Cycle 1
  TMZ 200 mg/m2 Day 1 - 5 Q4W PO Cycle 2 +
Drug: Cisplatin — Cisplatin 40 mg/m2 Q2W IV infusion Cycle 1 +
Drug: Nivolumab — Nivolumab 480 mg Q4W IV infusion Cycle 1 +

SUMMARY:
This study will test whether the combination of cisplatin, nivolumab, and temozolomide is an effective treatment for in people with advanced and/or metastatic colorectal cancer that is mismatch repair-proficient (MMR-proficient). The researchers will also look at how safe the study drug combination is in participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative is willing and able to provide written informed consent/assent for the trial.
* Histologically- or cytologically- confirmed colorectal adenocarcinoma.
* Locally advanced unresectable or metastatic CRC.
* Undergone testing for MSI/dMMR and determined to be MSS or MMR proficient.
* Undergone testing for BRAF and POLE and determined to be wild type.
* Subjects must be refractory to, or intolerant of, at least 2 lines of standard chemotherapy, according to NCCN guidelines for patients eligible for intensive therapy, or have received prior FOLFOXIRI. Patients are considered refractory if progressed within 3 months of last dose, or within 6 months of completing adjuvant FOLFOX/CAPEOX. At a minimum, such therapies should include oxaliplatin, irinotecan and a fluoropyrimidine.
* At least one index lesion which is measurable based on RECIST 1.1.
* Be ≥ 18 years of age on day of signing informed consent.
* Consent for use of archival tissue and blood draws for research purposes.
* Have an ECOG performance status of 0 or 1.
* Demonstrate adequate organ function as defined in Table 6.1, all screening labs should be performed within 28 days of treatment initiation.
* Adequate organ function, defined as:

  * Absolute Neutrophil Count ≥ 1,500/mcL.
  * Platelet count ≥ 100,000/mcL.
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥60 mL/min for subjects with creatinine levels >1.5 ULN.
  * WBC ≥ 2000/μL
  * Hemoglobin ≥ 9.0 g/dL
  * AST and ALT ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with liver metastases.
  * Bilirubin ≤ 1.5 × ULN or Direct bilirubin ≤ ULN for subjects with bilirubin levels >1.5
  * INR/PT and PTT ≤1.5 X ULN unless on anticoagulant therapy and PT/PTT within therapeutic range.

aCreatinine clearance should be calculated per institutional standard.

* Adequate method of contraception.

Exclusion Criteria:

* Subject is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg/day prednisone, or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Inhaled or topical steroids are permitted in the absence of active autoimmune disease
* Prior chemotherapy, targeted small molecule therapy, or biological therapy, within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (exc. alopecia).
* If subject received major surgery, they must have recovered adequately prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment.
* Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has an active, known or suspected autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy, type 1 diabetes mellitus are permitted. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or it is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months for females, 7 months for males after the last dose of trial treatment.
* Prior anti-PD-1, anti-PDL-1, anti-PDL-2, anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Subject is a prisoners, or compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Response | 1 year
  will be evaluated in this study using the new international criteria proposed in RECIST 1.1 [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor and the shortest diameter of malignant lymph nodes are used with the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm